CLINICAL TRIAL: NCT01701323
Title: Pilot Study Evaluating the Use of Ex Vivo Expanded Cord Blood Progenitors as Supportive Care Following Chemotherapy (FLAG) in Patients With AML or Acute Leukemia of Ambiguous Lineage
Brief Title: Expanded Cord Blood Cell Infusion Following Combination Chemotherapy in Younger Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Nohla Therapeutics, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2584; NCI-2012-01724 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2584; 2584.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Acute Leukemia of Ambiguous Lineage; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute | interventions — Cytarabine; Filgrastim; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Ex-vivo expanded cord blood progenitors) (Experimental): Patients receive filgrastim SC or IV on days 1-7, fludarabine phosphate IV QD over 30 minutes on days 2-6, cytarabine IV QD over 4 hours on days 2-6, and ex-vivo expanded cord blood progenitor cells IV over 30 minutes on day 8.
  Interventions: Biological: Ex-Vivo Expanded Cord Blood Progenitor Cell Infusion; Drug: Cytarabine; Drug: Filgrastim; Drug: Fludarabine Phosphate

INTERVENTIONS:
Biological: Ex-Vivo Expanded Cord Blood Progenitor Cell Infusion — Given IV
  Other Names: NLA101; Dilanubicel
Drug: Cytarabine — Given IV
Drug: Filgrastim — Given SC or IV
Drug: Fludarabine Phosphate — Given IV

SUMMARY:
This pilot clinical trial studies infusion of expanded cord blood hematopoietic progenitor cells following combination chemotherapy in treating younger patients with acute myeloid leukemia that has relapsed or has not responded to treatment. Chemotherapy drugs work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Chemotherapy also kills healthy infection-fighting cells, increasing the risk of infection. The infusion of expanded cord blood hematopoietic progenitor cells may be able to replace blood-forming cells that were destroyed by chemotherapy. This cellular therapy may decrease the risk of infection following chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of AML or acute leukemia of ambiguous lineage according to World Health Organization (WHO) classification with >= 5% of disease in bone marrow (BM)
* Recipients of prior allogeneic hematopoietic stem cell transplantation for AML or acute leukemia of ambiguous lineage are eligible if they do not have graft-versus-host disease (GVHD) or they have quiescent GVHD whether or not they are receiving immunosuppressive therapy
* Must have a Lansky or Karnofsky performance status of >= 50; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Patients must have recovered from the acute toxicity of all prior chemotherapy
* The following amounts of time must have elapsed prior to entry on study:

  * 2 weeks from local radiation therapy (XRT)
  * 8 weeks from prior craniospinal or if > 50% of the pelvis has been irradiated
  * 6 weeks must have elapsed if other bone marrow radiation has occurred
* Adequate cardiac, renal, pulmonary, and hepatic function
* Patient must have a life expectancy of at least 2 months
* Females of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Females of childbearing potential and males should agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation

Exclusion Criteria:

* Recipients of prior allogeneic hematopoietic stem cell transplant (HSCT) with active acute or chronic GVHD
* Patients with history of Down's syndrome, Fanconi anemia or other known marrow failure condition
* Patients currently receiving other investigational drugs are not eligible
* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol with the exception of intrathecal chemotherapy; this includes the tyrosine kinase inhibitor sorafenib which must not be initiated until patient demonstrates count recovery
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled despite appropriate antibiotics or other treatment; uncontrolled systemic infections require infectious disease consultation for verification
* Patients who are platelet refractory prior to initiation of protocol therapy
* Pregnant or lactating patients
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results

Ages: 6 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2012-12-10 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Incidence of NCI CTCAE grade > 3 infusional toxicities | Up to 2 years
Occurrence of transfusion associated graft versus host disease | Up to 2 years
Incidence of platelet refractoriness in the presence of alloimmunization as a direct result of ex vivo expanded cord blood product infusion | Up to 2 years
Incidence of delayed marrow recovery | Up to day 42
  Failure to achieve ANC >= 500 cells/µl by day 42 post treatment with marrow cellularity < 5% and marrow blast count < 5%.
Rate of treatment related mortality | Up to 2 years

SECONDARY OUTCOMES:
Time to neutrophil recovery | Up to 2 years
  ANC >= 100 cells/ul and 500 cells/ul
In vivo persistence of ex vivo expanded cellular therapy | Up to 2 years
  Assessed by peripheral blood cell sorted deoxyribonucleic acid (DNA) chimerisms of the cluster of differentiation myeloid and lymphoid cell lineages as well as whole marrow chimerisms.
Patient and infused expanded cord blood cells immune interaction | Up to 2 years
  Assessed by performing host-donor studies.
Incidence of NCI CTCAE grade 3 or 4 infections | First 30 days following FLAG administration
Incidence of NCI CTCAE grade > 3 chemotherapy-related toxicity in the first 30 days following fludarabine phosphate, cytarabine, and filgrastim (FLAG) therapy | First 30 days following FLAG administration
Rate of complete remission | Up to 2 years
Leukemia-free survival | Up to 2 years
Overall survival | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ann Dahlberg, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington